CLINICAL TRIAL: NCT00830050
Title: A Study To Determine The Ability Of FMRI To Detect And Quantify The Effect Of Naproxen On Osteoarthritis Of The Hand
Brief Title: Brain Imaging To Examine The Effect Of Naproxen In Hand Osteoarthritis Patients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: King's College London (Other)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: A9001399
Record Dates: First submitted 2009-01-26; First posted 2009-01-27 (Estimated); Last update posted 2011-03-14 (Estimated); Status verified 2011-03

CONDITIONS: Osteoarthritis
Keywords: fMRI functional magnetic resonance imaging Pain
MeSH Terms: conditions — Osteoarthritis | interventions — Naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Naproxen
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naproxen — 500 mg BID 7 days
  Arms: Arm 1
Drug: Placebo — BID 7 days
  Arms: Arm 2

SUMMARY:
The study hypothesis is that the relief of pain in patients with osteoarthritis in the hand can be detected by a form of brain scanning that detects which parts of the brain are activated when pain is felt.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed, post-menopausal female, any race, 50-80 years
* Clinical diagnosis of osteoarthritis of the hand
* Estimated pain in this joint of at least 5 on a scale of 0 to 10

Exclusion Criteria:

* Any patient who smokes more than 5 cigarettes per day
* Patients receiving some anti-depressant drugs unless the dose is stable
* Patients unable to be admitted or lie still in an MRI scanner

Ages: 50 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Changes in voxel-wise Blood Oxygen Level Dependent (BOLD) signal throughout the brain and changes in pre-defined brain regions of interest. | 22 days

SECONDARY OUTCOMES:
Whole brain resting-state distribution of Cerebral Blood Flow | 22 days
Psychometric measures of pain, namely Daily Pain Diaries and Present Pain Intensity | 22 days
Pain induced by a grip task measured with a Visual Analogue Scale (VAS), the Short-Form McGill Pain Questionnaire and patient-rated wrist/hand evaluation (PRWHE) | 22 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Denmark Hill, London, United Kingdom

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9001399&StudyName=Brain%20Imaging%20To%20Examine%20The%20Effect%20Of%20Naproxen%20In%20Hand%20Osteoarthritis%20Patients